CLINICAL TRIAL: NCT05845801
Title: Prospective Registry of Young-Adult Patients Diagnosed With Pancreatic Cancer
Acronym: PanC-YOUNG
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: 3968
Record Dates: First submitted 2023-04-07; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Registries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Register — Prospective collection of epidemiological, clinical, and pathological data of patients diagnosed with early-onset pancreatic cancer (EO-PDAC) - namely, individuals who have received a diagnosis of pancreatic cancer before, or at, the age of 55 years old.

SUMMARY:
The objective of the present registry is the creation of a prospective registry collecting clinico-pathological and genomic data, along with survival outcomes, of individuals diagnosed with PDAC at or before the age of 55 years old. This registry is intended with the aim of using collected data for future clinical trials, both prospective and retrospective.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤55 years old at the time of diagnosis of pancreatic cancer
* Age ≥ 18 years
* Written informed consent obtained.

Exclusion Criteria:

* Any pancreatic neoplasm other than pancreatic cancer (e.g. cholangiocarcinoma, ampullary cancer,duodenal cancer, non-invasive mucinous cystic neoplasm, pancreatic intra-epithelial neoplasia 1 and 2, non-invasive intraductal papillary mucinous neoplasm, serous cystic neoplasm, pseudo papillary solid tumor, neuroendocrine tumor)
* Absence of informed consent.
* Age < 18 years or > 55 years old at the time of diagnosis of pancreatic cancer

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: The target population is represented by individuals who have received a pathological diagnosis of pancreatic cancer before the age of 55 years old (namely, EO-PDAC patients). No subject will be financially compensated for their participation.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2052-09-30 (Estimated); Study Completion 2052-09-30 (Estimated)

PRIMARY OUTCOMES:
Register of young PDAC patients | 30 years
  Prospective collection of epidemiological, clinical, and pathological data of patients diagnosed with early-onset pancreatic cancer (EO-PDAC) - namely, individuals who have received a diagnosis of pancreatic cancer before, or at, the age of 55 years old.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided